CLINICAL TRIAL: NCT00170430
Title: Reducing Vaginal Infections in Women at Risk for HIV-1
Brief Title: Reducing Vaginal Infections in Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Dr. Scott McClelland, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20486-A; 01-0777-A 01 (Other: University of Washington Human Subjects Division); 02-125
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Bacterial Diseases; Other Mycoses; Sexually Transmitted Infection
Keywords: HIV-1, sexually transmitted diseases, females, Kenya
MeSH Terms: conditions — Bacterial Infections; Sexually Transmitted Diseases | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole
Drug: Metronizadole

SUMMARY:
The purpose of this study is to see if taking medication once a month can help to decrease the risk of vaginal infections. Additionally, researchers will study whether personal habits, such as douching, bathing, and sexual practices can influence the risk of vaginal infections. Vaginal infections may influence the risk of becoming infected with HIV-1 and other sexually transmitted diseases (STDs). Study participants will include 400 female prostitutes ages 16 and older, living in Mombasa. Study procedures will include sexual behavior questions, physical examinations including pelvic exams, testing of vaginal and cervical secretions for STDs, urine collection and blood samples. Participants will receive 2 different types of pills to treat vaginal infections (metronidazole or fluconazole) or placebo (contains no medication). Participants will be involved in study related procedures for 1 year and will return to the study clinic at one month intervals.

DETAILED DESCRIPTION:
Prospective studies in Africa have demonstrated that vaginal infections are associated with a significant increase in a woman's risk of infection with HIV-1. Further clinical and epidemiological research is needed to evaluate strategies for prevention and treatment of vaginal infections as a means of reducing HIV-1 acquisition. Developing a vaginal health intervention to reduce the risk of HIV-1 infection is a particularly important goal in sub-Saharan Africa, where female controlled strategies for reducing the risk of HIV-1 transmission may be an important means of decreasing the spread of the epidemic. This study will evaluate the efficacy of a regimen for reducing the rate of vaginal infections. The study is a double blind, randomized, controlled trial of monthly treatment with single-dose metronidazole and fluconazole as a means of decreasing vaginal infections and promoting normal vaginal flora in HIV-1 seronegative female sex workers (FSWs) in Mombasa, Kenya. Participants will be recruited from an existing cohort of HIV-1 seronegative FSWs followed at a municipal sexually transmitted disease (STD) clinic in Mombassa, Kenya, since February 1993. Participants will be randomized to treatment with metronidazole 2 grams plus fluconazole 150 mg once a month or placebo. All patients will be asked to return for follow-up after 1 month. All women in the study will be treated as indicated for symptomatic vaginal infections, other genital track infections and followed until they have completed 12 monthly follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Women who do not currently have symptoms of vaginal itching or discharge. Women with these symptoms may be treated and enrolled at a subsequent monthly visit when they are asymptomatic.
* Those who are currently menstruating may be enrolled after the completion of menses.

Exclusion Criteria:

* Pregnancy
* Lactation
* History of adverse reactions to the study medications
* Alcoholism or inability to abstain from alcohol for 48 hours following treatment
* Women who do not anticipate living in Mombasa for a year following enrollment.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 2003-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Scott McClelland, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Ganjoni Municipal Communicable Diseases Control Centre, Mombasa, Kenya